CLINICAL TRIAL: NCT03462108
Title: A Prospective Intervention Phase I Study in Three Age De-escalating Group to Assess the Safety and Immunogenicity of Rotavirus (Bio Farma) Vaccine in Adults, Children & Neonates
Brief Title: Safety and Immunogenicity of Rotavirus (Bio Farma) Vaccine in Adults, Children & Neonates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RV 0117
Record Dates: First submitted 2017-09-29; First posted 2018-03-12 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2018-04

CONDITIONS: Safety Issues
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Intervention Model Description: * Adults and Children Group: Experimental, open labeled, prospective intervention study
  * Neonates Group: Experimental, randomized, double blind, prospective intervention study
Who Masked: Participant, Investigator
Masking Description: The study for the neonates is double-blind, randomized study. While, the study for the adults and childrens is open-labeled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Rotavirus (Bio Farma) Vaccine-Adult (Experimental): 1 doses of 1 ml of Rotavirus vaccine per oral
  Interventions: Biological: Rotavirus (Bio Farma) Vaccine
- Rotavirus (Bio Farma) Vaccine-Children (Experimental): 1 doses of 1 ml of Rotavirus vaccine per oral
  Interventions: Biological: Rotavirus (Bio Farma) Vaccine
- Rotavirus (Bio Farma) Vaccine-Neonates (Experimental): 3 doses of 1 ml of Rotavirus vaccine per oral
  Interventions: Biological: Rotavirus (Bio Farma) Vaccine
- Placebo-Neonates (Placebo Comparator): 3 doses of 1 ml of Placebo (contains 30% sucrose in DMEM) per oral
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Rotavirus (Bio Farma) Vaccine — Rotavirus (Bio Farma) Vaccine
  Arms: Rotavirus (Bio Farma) Vaccine-Adult; Rotavirus (Bio Farma) Vaccine-Children; Rotavirus (Bio Farma) Vaccine-Neonates
Other: Placebo — Placebo contains 30% sucrose in DMEM
  Arms: Placebo-Neonates

SUMMARY:
This study is to assess the safety of Rotavirus (Bio Farma) vaccine in adults, children and neonates.

DETAILED DESCRIPTION:
To describe the safety of this vaccine after each immunization. To assess preliminary information of immunogenicity following Rotavirus (Bio Farma) vaccine immunization.

ELIGIBILITY:
Inclusion Criteria for Adults:

* Healthy Adults as determined by clinical judgment, including a medical history, physical exam and laboratory results, which confirms the absence of a current or past disease state considered significant by the investigator.
* Subjects have been informed properly regarding the study and signed the informed consent form.
* Subject will commit to comply with the instructions of the investigator and the schedule of the trial.

Inclusion Criteria for Children:

* Healthy Children as determined by clinical judgment, including a medical history and physical exam, which confirms the absence of a current or past disease state considered significant by the investigator.
* Parents/guardian(s) have been informed properly regarding the study and signed the informed consent form
* Parent/guardian(s) will commit to comply with the instructions of the investigator and the schedule of the trial.

Inclusion Criteria for Neonates:

* Neonate 0-5 days of age at the time of first dose, with cord blood available
* Neonate is in good health as determined by clinical judgment, including a medical history and physical exam, which confirms the absence of a current or past disease state considered significant by the investigator.
* The neonate was born full term (minimum of 36 completed weeks and maximum of 42 completed weeks gestation).
* Neonate birth weight 2500-4000 g inclusive.
* Parents or guardians have been informed properly regarding the study and signed the informed consent form
* Parents or guardians will commit to comply with the instructions of the investigator and the schedule of the trial

Exclusion Criteria for Adults:

* Subject concomitantly enrolled or scheduled to be enrolled in another trial
* Any direct relatives relationship with the study team.
* Evolving mild, moderate or severe illness, especially infectious diseases or fever (axillary temperature ³ 37.5°C) within the 48 hours preceding enrollment.
* Known history of allergy to any component of the vaccines
* Known history of immunodeficiency disorder (HIV infection, leukemia, lymphoma, or malignancy)
* Gastroenteritis in the 24 hours preceding enrollment.
* History of uncontrolled coagulopathy or blood disorders contraindicating for phlebotomy.
* Subject who has received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products, or corticosteroid therapy and other immunosuppresant).
* Subject consuming or expect to consume a probiotics within one week before and after vaccination
* Any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objectives.
* Pregnancy & lactation (Adults).
* Subject already immunized with any vaccine within 4 weeks prior and expects to receive other vaccines within 4 weeks following immunization.
* Subject planning to move from the study area before the end of study period.

Exclusion Criteria for Children:

* Subject concomitantly enrolled or scheduled to be enrolled in another trial
* Any direct relatives relationship with the study team
* Evolving mild, moderate or severe illness, especially infectious diseases or fever (axillary temperature ³ 37.5°C ) within the 48 hours preceding enrollment
* Known history of allergy to any component of the vaccines
* Known history of immunodeficiency disorder (HIV infection, leukemia, lymphoma, or malignancy)
* Gastroenteritis in the 24 hours preceding enrollment.
* Any clinically significant history of chronic gastrointestinal disease including uncorrected congenital malformation of gastrointestinal tract that would predispose for Intusussception.
* History of uncontrolled coagulopathy or blood disorders contraindicating for phlebotomy.
* Subject who has received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products or corticosteroid therapy and other immunosuppresant).
* Subjects consuming or expect to consume a probiotics within one week before and after vaccination.
* Any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objectives.
* Individuals who have previously received any rotavirus vaccine.
* Subject already immunized with any vaccine within 4 weeks prior and expects to receive other vaccines within 4 weeks following immunization.
* Subject planning to move from the study area before the end of study period

Exclusion Criteria for Neonates:

* Subject concomitantly enrolled or scheduled to be enrolled in another trial.
* Any direct relatives relationship with the study team.
* Evolving mild, moderate or severe illness, especially infectious diseases or fever (axillary temperature ³ 37.5°C) within the 48 hours preceding enrollment.
* Subject with known or suspected history of allergy to any component of the vaccines.
* Subject with a biological mother with a known or suspected human immunodeficiency virus (HIV) infection.
* Subject with known or suspected major congenital malformations or genetically determined disease.
* Subject with intussusception.
* Subject with a known or suspected disease of uncontrolled coagulopathy or blood disorders contraindicating for phlebotomy.
* Subject with a known or suspected disease of the immune system or those who has received immunosuppresive therapy, including immunosuppresive courses of systemic corticosteroid.
* Subject who have ever received any blood products, including immunoglobulin, or for whom receipt of any blood product during the course of study.
* Any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objectives.
* Subject immunized with non- EPI vaccines.
* Gastroenteritis in the 24 hours preceding enrollment.
* Subject planning to move from the study area before the end of study period.

Ages: 1 Minute to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Solicited symptoms after each immunization | 0-7 days
  Number of subjects with solicited systemic and gastrointestinal symptoms in the day 0-7 following each dose of investigational product

SECONDARY OUTCOMES:
Adverse events of Rotavirus (Bio Farma) vaccine | 28 days
  Number and percentage of subjects with unsolicited Adverse Events (AE) in the day 0-28 following each dose of investigational product
Serious adverse events of Rotavirus (Bio Farma) vaccine | 28 days
  Number and percentage of subjects with Serious Adverse Events (SAE) within 28 days after each dose of investigational product
Adverse events of Rotavirus (Bio Farma) vaccine compare to placebo in neonates group | 28 days
  Number and percentage of subject with adverse event (AE) within 28 days after each dose of investigational product compare to placebo (in neonates group)
Serious adverse events of Rotavirus (Bio Farma) vaccine compare to placebo in neonates group | 28 days
  Number and percentage of subject with Serious Adverse Events (SAE) within 28 days after each dose of investigational product compare to placebo (in neonates group)
Number of subject who has abnormality value of routine hematology and biochemical evaluation that probably related to the vaccination | 7 days
  Deviation in routine hematology and biochemical evaluation
Excretion of rotavirus in stools in neonates group | 3-7 days
  Number of neonates with rotavirus excretion in stools
Number of subjects with >=3 times increasing antibody from baseline to post investigational product dosing | 4-6 weeks after last immunization
  Subjects with >=3 times increasing antibody from baseline to post investigational product dosing
Serum anti-rotavirus immunoglobulin (Ig)A following immunization | 4-6 weeks after last immunization
  Serum anti-rotavirus immunoglobulin (Ig)A before and after last immunization
Serum neutralizing antibody (SNA) following immunization | 4-6 weeks after last immunization
  Serum neutralizing antibody (SNA) before and after last immunization
Geometric Mean Titer (GMT) following immunization | 4-6 weeks after last immunization
  Geometric mean titer (GMT) before and after last immunization

CONTACTS AND LOCATIONS:
Overall Officials: Jarir At Thobari, Principal Investigator — Pediatric Research Office (PRO), Departemen Ilmu Kesehatan Anak, Fakultas Kedokteran UGM/RSUP Dr. Sardjito
Locations (4):
- Indonesia (4):
  - Gantiwarno Primary Health Center, Klaten, Central Java
  - Klaten Selatan Primary Health Center, Klaten, Central Java
  - Ngawen Primary Health Center, Klaten, Central Java
  - RS Soeradji Tritonegoro, Klaten, Central Java

IPD SHARING:
Plan to Share IPD: No